CLINICAL TRIAL: NCT06572787
Title: Evaluation of Family Centered Service in the Physiotherapy and Rehabilitation Processes of Children with Cerebral Palsy
Brief Title: Family Centered Services in Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mustafa Ocalan, Principal Investigator, Hacettepe University
Other Study IDs: HACETTEPEU-SBF-MO-01
Record Dates: First submitted 2024-08-22; First posted 2024-08-27 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-08

CONDITIONS: Cerebral Palsy
Keywords: Physiotherapy; Rehabilitation; Family Centered Services; Impact Family; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
To examine the family-centered service characteristics of physiotherapy and rehabilitation services received by children with cerebral palsy (CP) and to investigate the affecting factors.

DETAILED DESCRIPTION:
Children with Cerebral Palsy (CP) attend special education and rehabilitation centers to receive physiotherapy and rehabilitation (PT) services, and it is very important for parents to be informed about the services offered in these centers. Our aim in the study was to examine which factors affect family-centered characteristics and parental perceptions in the PT services received by children with CP. For this purpose, 100 children diagnosed with CP between the ages of 2-18 and their parents were included in the study. The Measure of Processes Care (MPOC) survey was used to assess parents' perceptions of the family-centered features of (PT) services. These perceptions were examined to determine whether they vary depending on the child's age, functional level, parents' educational status, the impact of their disabled children, and health-related quality of life. The Family Impact Scale was used to measure parents' level of influence from their disabled children, and the Nottingham Health Profile survey was used to evaluate their health-related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Having a child aged between 2 and 18 years diagnosed with cerebral palsy
* Receiving physiotherapy and rehabilitation services for at least one year
* The family's consent to participate in the study and their approval for their child to be assessed by the researcher physiotherapist and for their information to be collected within the scope of the study

Exclusion Criteria:

* Parents over the age of 65
* Parents who do not speak Turkish
* Having another child with a disability

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with cerebral palsy between the ages of 2 and 18 who have received physiotherapy and rehabilitation services for at least one year and their parents
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
Measure of Processus of Care | 3 months
  Measure of Processus of Care-20 (MPOC-20) survey was administered to assess parents' perceptions of the family-centered features of physiotherapy and rehabilitation services. The appropriate answers to the questions in the survey are marked with a number from 1 (strongly disagree) to 7 (strongly agree). A value of zero (0) indicated not personally relevant.

SECONDARY OUTCOMES:
Impact on Family Scale | 3 months
  The Impact on Family of Scale (IPFAM) scale was used to determine impact of the child with CP on parents. IPFAM consists of 33 items in total. The family's level of involvement is measured under 5 headings.The scale has a Likert-type evaluation ranging from 1 to 4. A low score from the survey indicates a high level of family involvement
Nottingham Health Profile | 3 months
  The Nottingham Health Profile (NHP) was used to measure parents' health-related quality of life. NHP is a scale used to assess quality of life. This profile was developed to measure the physical, emotional and social health status of individuals. The questionnaire consists of 7 subsections and a total of 45 items. The maximum score that can be obtained from the questionnaire is 607. High scores indicate low quality of life and low scores indicate high quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Öcalan, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe Universty, Ankara, Sıhhiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No